CLINICAL TRIAL: NCT05531032
Title: Health-related Quality of Life Following Extracorporeal Membrane Oxygenation Due to Coronavirus Disease 2019.
Brief Title: HRQOL of Life After ECMO Due to COVID-19.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Martina Hermann, Principal investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2440/2020
Record Dates: First submitted 2022-08-30; First posted 2022-09-07 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-11

CONDITIONS: ARDS; COVID-19 Pneumonia; Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Intervention Model Description: Phone Interview
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Phone Interview — Phone interview questionnaire

SUMMARY:
We intend to prospectively investigate physical and mental state (HRQOL) by means of quantitative telephone interviews after hospital discharge in patients surviving COVID-19 ARDS and ECMO therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients surviving COVID-19 ARDS and ECMO therapy

Exclusion Criteria:

* no consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 44 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
HRQOL after COVID-19 ARDS and ECMO therapy | 1 year
  Health-related quality of life will be delineated by means of a quantitative questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hermann, Dr., Principal Investigator — MUW
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol